CLINICAL TRIAL: NCT05536232
Title: Residual Insulin Secretion in Patients With Type 1 Diabetes Under a Low Carbohydrate Diet or a Ketogenic Diet
Acronym: KetoDiab
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: APHP211325; 2022-A00523-40 (Registry Identifier: DRCB)
Record Dates: First submitted 2022-09-07; First posted 2022-09-10 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2022-06

CONDITIONS: Type1 Diabetes
Keywords: type 1 diabetes; low carbohydrate diet; ketogenic diet
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Diet, Carbohydrate-Restricted

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LCD (Experimental)
  Interventions: Behavioral: Low carbohydrate diet

INTERVENTIONS:
Behavioral: Low carbohydrate diet — Low carbohydrate diet under 75 g per day

SUMMARY:
Low Carbohydrate Diet (LCD) (< 130 g of carbohydrate per day) and ketogenic diet (< 50 g of carbohydrate per day) are popular among patients with type 1 diabetes (T1D). In most cases, LCD allow a better glycemic control and a important decrease of insulin requirements that cannot, however, be the sole result of low carbohydrate intake. However, due to the increase production of ketone bodies and the decrease of the insulin/glucagon rate, this diet is not without risk in T1D patients and some of them develop ketoacidosis.

Type 1 diabetes is a autoimmune disease defined by the destruction of the pancreatic beta cells by the effector T cells, in condition of low regulatory T cells (Tregs). Indeed, some nutrients could regulate the plasticity and the function of Tregs, and be involved in the control of some autoimmune diseases in animals models thanks to a direct effect on immune cells of the digestive tract or an indirect effect by microbiota modulation.

The study hypothesises that LCD may be able to restore residual insulin secretion in some patients by modulating immunity. The metabolic mechanisms leading to the effects described in patients with T1D patients under LCD have not been studied : in particular, there is no data on the evolution of the residual insulin secretion and no immunological parameter has been studied on these patients.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older
* type 1 diabetes for less than 20 years
* willing to start a low carbohydrate diet of less than 75 g per day
* under continuous glucose monitoring
* having been informed about the study and having given their written and informed consent

Exclusion Criteria:

* already on a low carbohydrate diet of less than 100 g per day
* history of ketoacidosis within the last 5 years, except during diabetes diagnosis
* autoimmune disease, except thyroiditis
* immunosuppressive treatment
* hepatitis B virus, hepatitis C virus or human immunodeficiency virus infection
* ongoing cancer or history of cancer within the past 5 years, except in situ cervical cancer or basal cell cancer with early treatment
* participation to another interventional study within the past 3 months
* pregnancy or breast feeding
* no affiliation to a social security scheme
* patients subject to legal protection measures
* unability to give consent for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-10-17 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Peptide C evolution | Day 0 and day 90
  Measure of the area under the curve of the peptide C dosage

SECONDARY OUTCOMES:
HbA1C measure | Day 0 and day 90
Insulin-dose adjusted A1c (IDAA1C) index calculation | Day 0 and day 90
Weight measure | Day 0 and day 90
Fat mass percentage measure | Day 0 and day 90
Lean mass percentage measure | Day 0 and day 90
Daily dose of insulin | Every day from day 0 to day 90
Circulating rate of Tregs | Day 0 and day 90
Circulating rate of cytokines | Day 0 and day 90

CONTACTS AND LOCATIONS:
Locations (1):
- AP-HP - Pitié-Salpêtrière Hospital, Paris, France